CLINICAL TRIAL: NCT07358065
Title: Clinical Application of Dynamic Multimodal Analgesia Regimen After Perianal Abscess Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Principal Investigator, Hong Wu, Supervisory assistant of Scientific Research Department, The Affiliated Hospital of Putian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PutianU-014
Record Dates: First submitted 2026-01-03; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Clinical Application of Dynamic Multimodal Analgesia Regimen After Perianal Abscess Surgery
Keywords: Perianal Abscess; Postoperative Pain; Dynamic Assessment; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A ：Conventional Analgesia Group (Other): Adopts the traditional analgesic mode.
  Interventions: Drug: the traditional analgesic mode
- Group B：Western Medicine Multimodal Analgesia Group (Other): Implements a dynamic assessment-based full-course multimodal analgesia strategy.
  Interventions: Behavioral: Western Medicine Multimodal Analgesia
- Group C：Integrated Traditional Chinese and Western Medicine Multimodal Analgesia Group (Other): Integrates characteristic traditional Chinese medicine nursing interventions on the basis of western medicine multimodal analgesia.
  Interventions: Behavioral: Integrated Traditional Chinese and Western Medicine Multimodal Analgesia

INTERVENTIONS:
Drug: the traditional analgesic mode — Adopt the traditional analgesic mode: conduct NRS assessment and intervention only when the patient takes the initiative to complain of pain, without fixed assessment time points. Intervene when the pain score is ≥4 points, and no prophylactic medication is administered. Medication use refers to the conventional plan (e.g., flurbiprofen injection, diclofenac sodium capsules, etc.).
  Arms: Group A ：Conventional Analgesia Group
Behavioral: Western Medicine Multimodal Analgesia — Collect baseline NRS score 24 hours before surgery. After surgery, assess NRS in resting and active states at fixed daily time points (e.g., 08:00, 16:00), and conduct on-demand assessment for breakthrough pain. Reassess during outpatient follow-up at 2 weeks and 1 month after discharge.
  1. Stepwise medication intervention: Administer medications in a stepwise manner based on NRS score. For scores ≤3 points, prioritize non-pharmacological interventions; for scores ≥4 points, initiate NSAIDs, acetaminophen, etc.; for moderate to severe pain, administer bucinazine, pethidine, or other medications as needed.
  2. Non-pharmacological auxiliary measures: Include potassium permanganate sitz bath, health education, psychological counseling, etc.
  3. Dynamic adjustment: The pain management team conducts daily rounds to individually adjust the plan based on assessment results.
  Arms: Group B：Western Medicine Multimodal Analgesia Group
Behavioral: Integrated Traditional Chinese and Western Medicine Multimodal Analgesia — On the basis of western medicine multimodal analgesia, integrate characteristic traditional Chinese medicine nursing interventions, such as auricular point pressing, wrist-ankle acupuncture, traditional Chinese medicine sitz bath, etc.
  Arms: Group C：Integrated Traditional Chinese and Western Medicine Multimodal Analgesia Group

SUMMARY:
This study aims to investigate whether the full-course multimodal analgesia regimen based on dynamic assessment (including the integrated traditional Chinese and Western medicine mode) can alleviate postoperative pain, reduce opioid dosage, and decrease the incidence of complications in patients with perianal abscess. It also intends to verify the clinical advantages of the integrated traditional Chinese and Western medicine multimodal regimen and establish a promotable standardized pain management pathway. A total of 135 eligible patients will be enrolled and divided into three groups in a 1:1:1 ratio using a single-center, prospective, randomized parallel-controlled design. The specific grouping and intervention methods are as follows: ① Control Group (Group A): Adopts the traditional analgesic mode, where NRS assessment and intervention are conducted only when the patient actively complains of pain (medication administered for scores ≥4 points) without preemptive medication. Medications refer to conventional schemes (e.g., flurbiprofen, diclofenac sodium, etc.). ② Western Medicine Multimodal Analgesia Group (Group B): Implements dynamic assessment + stepwise medication intervention + non-pharmacological auxiliary measures. Baseline NRS score is collected 24 hours before surgery; pain at rest and during activity is assessed at fixed time points after surgery; NSAIDs, opioids, and other medications are administered as needed, combined with potassium permanganate sitz bath, health education, etc. ③ Integrated Traditional Chinese and Western Medicine Multimodal Analgesia Group (Group C): Integrates characteristic traditional Chinese medicine nursing interventions (including auricular point pressing, wrist-ankle acupuncture, traditional Chinese medicine sitz bath, etc.) on the basis of Group B's intervention.

To evaluate the clinical efficacy of the dynamic multimodal analgesia regimen, this study will compare the following indicators among the three groups: NRS pain scores on postoperative days 1, 2, 3, 4, 5, as well as 2 weeks and 1 month after discharge; total postoperative analgesic consumption converted to morphine equivalent dose (MEDD); quality of life score assessed by the SF-36 scale; incidence of complications (such as urinary retention, secondary hemorrhage, etc.); sexual function recovery (assessed by the IIEF-5 scale for males and the FSFI scale for females); and patient satisfaction and compliance. The primary research hypothesis is: compared with conventional analgesia and western medicine-only multimodal analgesia, the integrated traditional Chinese and Western medicine multimodal analgesia regimen can significantly reduce patients' postoperative pain scores, decrease opioid dosage, improve quality of life and patient satisfaction, lower the incidence of complications, and enhance patients' sexual function recovery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary perianal abscess by clinical examinations (digital rectal examination, ultrasound, or MRI) and undergoing incision and drainage or radical surgical treatment;
* Abscess diameter ≥ 2 cm or accompanied by obvious abscess cavity formation;
* Patients are willing and able to participate in the pain management plan, understand the importance of pain management, and actively cooperate;
* No severe coagulation disorders.

Exclusion Criteria:

* Complicated with specific infectious diseases such as Crohn's disease or tuberculosis;
* Unclear source of postoperative pain (i.e., the patient's pain is uncertain or unrelated to the surgery);
* Having definite contraindications, including drug allergies or inability to accept certain pain management methods adopted in the study;
* Pregnant or lactating women;
* Patients unable to cooperate with the study, such as those with cognitive impairment, history of mental illness, or communication difficulties;
* Patients with long-term use of analgesic drugs and developed drug tolerance;
* Complicated with uncontrolled cardiovascular and cerebrovascular diseases (NYHA cardiac function Class Ⅲ-Ⅳ), liver or kidney insufficiency (Child-Pugh Class C or eGFR < 30 ml/min/1.73m²), etc.;
* Abscess secondary to rectal tumors, trauma, or iatrogenic injury;
* Postoperative occurrence of severe complications (e.g., massive hemorrhage, sepsis) or combined infection in other parts;
* Patients receiving only non-surgical treatments such as simple puncture and aspiration of pus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | From enrollment to 1 month after discharge
  Postoperative pain score (NRS，Numeric Rating Scale): Record pain scores at rest and during activity on postoperative days 1, 2, 3, 4, 5, as well as at 2 weeks and 1 month after discharge, serving as the core assessment of the analgesic effect of the regimen.NRS，0 points indicate no pain, while 10 points represent the most severe pain.

SECONDARY OUTCOMES:
Secondary Efficacy Indicators | From enrollment to 1 month after discharge
  Total postoperative analgesic consumption: Convert all analgesics to morphine equivalent dose (MEDD) for intergroup comparison to evaluate the opioid-sparing effect of the regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Putian University, Putian, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Based on a strict commitment to participant privacy protection, compliance with the terms of the ethical review protocol, and adherence to the sponsoring institution's policies, IPD from this study will not be shared at this time.